CLINICAL TRIAL: NCT01385566
Title: A Partially Blinded Randomized Clinical Trial to Study the Immunogenicity and Safety of Intradermal Administration of ZOSTAVAX™ (V211)
Brief Title: A Study of Intradermal Administration of ZOSTAVAX™ (V211-051 AM2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V211-051
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Full Dose Subcutaneous (Active Comparator): Participants will receive a full dose of ZOSTAVAX™ administered subcutaneously on Day 1 of the study. Nine participants in this group will also receive saline placebo intradermally in the alternate limb on Day 1.
  Interventions: Biological: ZOSTAVAX™ (Zoster Vaccine Live) Full Dose Subcutaneous; Biological: Intradermal Placebo
- 1/3 Dose Subcutaneous (Experimental): Participants will receive a 1/3 dose of ZOSTAVAX™ administered subcutaneously on Day 1 of the study. Six participants in this group will also receive saline placebo intradermally in the alternate limb on Day 1. Participants will have the option to receive a full subcutaneous dose of ZOSTAVAX™ after completion of the study.
  Interventions: Biological: ZOSTAVAX™ (Zoster Vaccine Live) 1/3 Dose Subcutaneous; Biological: Intradermal Placebo
- Full Dose Intradermal (Experimental): Participants will receive a full dose of ZOSTAVAX™ administered intradermally on Day 1 of the study. Six participants in this group will also receive saline placebo intradermally in the alternate limb on Day 1. Participants will have the option to receive a full subcutaneous dose of ZOSTAVAX™ after completion of the study.
  Interventions: Biological: ZOSTAVAX™ (Zoster Vaccine Live) Full Dose Intradermal; Biological: Full Dose Intradermal Placebo
- 1/3 Dose Intradermal (Experimental): Participants will receive a 1/3 dose of ZOSTAVAX™ administered intradermally on Day 1 of the study. Six participants in this group will also receive saline placebo intradermally in the alternate limb on Day 1. Participants will have the option to receive a full subcutaneous dose of ZOSTAVAX™ after completion of the study.
  Interventions: Biological: ZOSTAVAX™ (Zoster Vaccine Live) Partial Doses Intradermal; Biological: Intradermal Placebo
- 1/10 Dose Intradermal (Experimental): Participants will receive a 1/10 dose of ZOSTAVAX™ administered intradermally on Day 1 of the study. Six participants in this group will also receive saline placebo intradermally in the alternate limb on Day 1. Participants will have the option to receive a full subcutaneous dose of ZOSTAVAX™ after completion of the study.
  Interventions: Biological: ZOSTAVAX™ (Zoster Vaccine Live) Partial Doses Intradermal; Biological: Intradermal Placebo
- 1/27 Dose Intradermal (Experimental): Participants will receive a 1/27 dose of ZOSTAVAX™ administered intradermally on Day 1 of the study. Six participants in this group will also receive saline placebo intradermally in the alternate limb on Day 1. Participants will have the option to receive a full subcutaneous dose of ZOSTAVAX™ after completion of the study.
  Interventions: Biological: ZOSTAVAX™ (Zoster Vaccine Live) Partial Doses Intradermal; Biological: Intradermal Placebo

INTERVENTIONS:
Biological: ZOSTAVAX™ (Zoster Vaccine Live) Full Dose Subcutaneous — One 0.65 mL injection subcutaneously on Day 1
  Other Names: V211
  Arms: Full Dose Subcutaneous
Biological: ZOSTAVAX™ (Zoster Vaccine Live) 1/3 Dose Subcutaneous — One approximately 0.22 mL injection subcutaneously on Day 1
  Other Names: V211
  Arms: 1/3 Dose Subcutaneous
Biological: ZOSTAVAX™ (Zoster Vaccine Live) Full Dose Intradermal — Two intradermal injections of approximately 0.15 mL each on Day 1
  Other Names: V211
  Arms: Full Dose Intradermal
Biological: ZOSTAVAX™ (Zoster Vaccine Live) Partial Doses Intradermal — One intradermal injection of approximately 0.1 mL on Day 1
  Other Names: V211
  Arms: 1/10 Dose Intradermal; 1/27 Dose Intradermal; 1/3 Dose Intradermal
Biological: Full Dose Intradermal Placebo — Two intradermal placebo injections of approximately 0.15 mL each on Day 1
  Arms: Full Dose Intradermal
Biological: Intradermal Placebo — One intradermal placebo injection of approximately 0.1 mL on Day 1
  Arms: 1/10 Dose Intradermal; 1/27 Dose Intradermal; 1/3 Dose Intradermal; 1/3 Dose Subcutaneous; Full Dose Subcutaneous

SUMMARY:
This study will compare the safety and immunogenicity of ZOSTAVAX™ (V211) administered both intradermally and subcutaneously at various doses.

DETAILED DESCRIPTION:
This is an exploratory, randomized, partially blinded, multicenter clinical study designed to compare safety and biomarkers of varicella zoster virus immunogenicity when administering ZOSTAVAX™ (V211) at various doses both intradermally and subcutaneously in healthy male and female participants 50 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

* Prior history of varicella (chickenpox) or residence in a country with endemic varicella zoster virus infection for at least 30 years
* Temperature less than 100.4 °F on day of vaccination
* Female participants of reproductive potential must have a negative pregnancy test and agree to remain abstinent or use two acceptable contraceptive methods for 3 months postvaccination
* In good health

Exclusion Criteria:

* History of hypersensitivity reaction to any vaccine component, including gelatin or neomycin
* Household exposure to pregnant women who have not had chickenpox and have not been vaccinated against varicella or to immunosuppressed/immunodeficient individuals
* Household or workplace exposure to children 18 months and younger who have not been vaccinated against varicella
* Prior history of herpes zoster
* Prior receipt of any varicella or zoster vaccine
* Received or is expected to receive immune globulin and/or blood products from 5 months prior to randomization through 42 days after vaccination
* On immunosuppressive therapy
* Known or suspected immune dysfunction
* Received a live virus vaccine or is scheduled to receive a live virus vaccine from 4 weeks prior to study vaccination through the completion of all study visits
* Received any inactivated vaccine or is scheduled to receive any inactivated vaccine from 7 days prior to study vaccination through 7 days postvaccination, except for inactivated influenza vaccine
* Not ambulatory
* Pregnant or breastfeeding
* Use of nontopical antiviral therapy with activity against herpes viruses
* Active untreated tuberculosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

REFERENCES:
- [Result] Beals CR, Railkar RA, Schaeffer AK, Levin Y, Kochba E, Meyer BK, Evans RK, Sheldon EA, Lasseter K, Lang N, Weinberg A, Canniff J, Levin MJ. Immune response and reactogenicity of intradermal administration versus subcutaneous administration of varicella-zoster virus vaccine: an exploratory, randomised, partly blinded trial. Lancet Infect Dis. 2016 Aug;16(8):915-22. doi: 10.1016/S1473-3099(16)00133-X. Epub 2016 Apr 6. PMID 27061887

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal
Started | 52 | 34 | 34 | 35 | 34 | 34
Completed | 51 | 34 | 34 | 34 | 34 | 34
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal | Total
Number analyzed (Participants) | 52 | 34 | 34 | 35 | 34 | 34 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (7.7) | 60.5 (7.5) | 62.1 (8.5) | 61.2 (8.7) | 61.6 (8.1) | 60.1 (7.1) | 60.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 17 | 17 | 16 | 24 | 125
  Male | 21 | 14 | 17 | 18 | 18 | 10 | 98

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Change From Baseline in Varicella Zoster Virus (VZV)-Specific Antibodies
Description: VZV antibody titers were measured by glycoprotein enzyme-linked immunosorbent assay at baseline and at 6 weeks after vaccine administration. The geometric mean fold change represents the 6-week value / the baseline value.
Time Frame: Baseline and 6 weeks following vaccine administration
Population: The population analyzed included participants who received vaccination and did not have any protocol deviations that may have interfered with the immune response.
Measure: Geometric Mean (90% Confidence Interval); unit: Geometric mean fold change
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal
Number analyzed (Participants) | 52 | 34 | 34 | 35 | 34 | 34
Geometric mean fold change | 1.74 [1.48 to 2.05] | 1.64 [1.35 to 2.00] | 3.24 [2.66 to 3.94] | 2.45 [2.02 to 2.97] | 2.21 [1.82 to 2.69] | 1.64 [1.35 to 2.00]

2. Primary Outcome: Number of Participants Reporting an Adverse Experience (AE)
Description: An AE is defined as any unfavorable and unintended change in the
  structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse experience.
Time Frame: Up to 42 days following vaccine administration
Population: The population analyzed was all randomized participants who received study vaccination
Measure: Number; unit: participants
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal
Number analyzed (Participants) | 52 | 34 | 34 | 35 | 34 | 34
participants | 30 | 10 | 27 | 23 | 21 | 19

3. Primary Outcome: Number of Participants Reporting a Serious Adverse Experience (SAE)
Description: An SAE is any adverse experience that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in or prolongs an existing inpatient hospitalization, is a congenital anomaly/birth defect in offspring of a study participant, is a cancer, or is another important medical event when, based on appropriate medical judgment, the event may jeopardize the participant and may require medical or surgical intervention.
Time Frame: Up to 42 days following vaccine administration
Population: The population analyzed was all randomized participants who received study vaccination
Measure: Number; unit: participants
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal
Number analyzed (Participants) | 52 | 34 | 34 | 35 | 34 | 34
participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Reporting a Serious Adverse Experience
Description: as for outcome 3
Time Frame: Within 5 days after the blood draw at approximately 20 months following vaccine administration
Population: The population analyzed was all randomized participants who received study vaccination and had a Month 20 visit and follow-up
Measure: Number; unit: Participants
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal
Number analyzed (Participants) | 22 | 16 | 10 | 13 | 15 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Reporting Specific Local Injection-site Adverse Experiences Prompted for on the Vaccine Report Card (VRC)
Description: The VRC actively prompts for local injection-site AEs of redness, swelling, and pain/tenderness and for the size of local injection-site reactions of redness and swelling that occur within 5 days of vaccination. The presence of varicella/varicella-like rash and herpes zoster/herpes zoster-like rash is also captured on the VRC. Participants receiving an injection in both limbs will be instructed to complete injection-site reaction information for each limb. All injection-site AEs were reported for the limb in which they occurred: V211 vaccine or placebo.
Time Frame: Up to 5 days following vaccine administration
Population: The population analyzed was all randomized participants who received study vaccination
Measure: Number; unit: Participants
Groups:
- Placebo: On Day 1 of the study, participants will receive a dose of ZOSTAVAX™ administered in one limb according to their randomized treatment group, and a dose of saline placebo in the alternate limb. Participants in this group were included in the analyses for the V211 treatment groups, and are replicated here specifically to report injection-site adverse experiences reported for the limb receiving a placebo injection.
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal | Placebo
Number analyzed (Participants) | 52 | 34 | 34 | 35 | 34 | 34 | 39
Participants
  Any injection-site AE | 27 | 7 | 27 | 22 | 19 | 19 | 5
  Injection-site anaesthesia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Injection-site erythema | 16 | 5 | 26 | 20 | 16 | 18 | 4
  Injection-site haematoma | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Injection-site induration | 5 | 2 | 12 | 12 | 11 | 10 | 1
  Injection-site pain | 15 | 5 | 8 | 9 | 5 | 6 | 0
  Injection-site pruritus | 1 | 2 | 3 | 3 | 1 | 1 | 0
  Injection-site rash | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Injection-site scab | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Injection-site swelling | 13 | 4 | 13 | 8 | 6 | 7 | 2

6. Primary Outcome: Number of Participants Reporting Systemic Adverse Experiences
Description: Systemic AEs included all reported AEs except injection-site AEs
Time Frame: Up to 42 days following vaccine administration
Population: The population analyzed was all randomized participants who received study vaccination
Measure: Number; unit: participants
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal
Number analyzed (Participants) | 52 | 34 | 34 | 35 | 34 | 34
participants | 12 | 6 | 6 | 4 | 5 | 6

7. Primary Outcome: Number of Participants Reporting a Non-injection-site Rash (Varicella, Varicella-like, Herpes Zoster, or Herpes Zoster-like)
Description: Non-injection-site rashes were examined by a study physician. Rashes suspected to be varicella/varicella-like or herpes zoster/herpes zoster-like were sampled for verification by polymerase chain reaction.
Time Frame: Up to 42 days following vaccine administration
Population: The population analyzed was all randomized participants who received study vaccination
Measure: Number; unit: participants
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal
Number analyzed (Participants) | 52 | 34 | 34 | 35 | 34 | 34
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were collected up to 20 months following vaccine administration. Other Adverse Events were collected up to 84 days following vaccine administration.
Description: Systemic adverse events are reported by V211 treatment group only. Injection-site adverse events are reported by V211 treatment group and placebo, according to the limb receiving the injection: V211 treatment or placebo.
Groups:
- Placebo: On Day 1 of the study, participants will receive a dose of ZOSTAVAX™ administered in one limb according to their randomized treatment group, and a dose of saline placebo in the alternate limb. Only injection-site adverse events occurring in the placebo limb are reported; systemic adverse events are reported by V211 treatment group only.
Arm/Group | Full Dose Subcutaneous | 1/3 Dose Subcutaneous | Full Dose Intradermal | 1/3 Dose Intradermal | 1/10 Dose Intradermal | 1/27 Dose Intradermal | Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/34 | 0/34 | 0/35 | 0/34 | 0/34 | 0/39
Other Adverse Events (participants affected / at risk) | 30/52 | 10/34 | 27/34 | 23/35 | 21/34 | 19/34 | 5/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Full Dose Subcutaneous (N=52) | 1/3 Dose Subcutaneous (N=34) | Full Dose Intradermal (N=34) | 1/3 Dose Intradermal (N=35) | 1/10 Dose Intradermal (N=34) | 1/27 Dose Intradermal (N=34) | Placebo (N=39)
Injection site erythema (General disorders) | 16 (25) | 5 (13) | 26 (58) | 21 (39) | 16 (20) | 18 (24) | 4 (10)
Injection site induration (General disorders) | 5 (9) | 2 (5) | 12 (17) | 12 (23) | 11 (11) | 10 (13) | 1 (1)
Injection site pain (General disorders) | 15 (15) | 5 (6) | 8 (17) | 9 (10) | 5 (5) | 6 (8) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 2 (4) | 4 (6) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 13 (23) | 4 (10) | 13 (33) | 8 (12) | 6 (6) | 7 (10) | 2 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0/0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0/0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication or presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.